CLINICAL TRIAL: NCT05340907
Title: Patient Satisfaction and Tolerability Using Virtual Reality (VR) as Adjunctive Treatment During Flexible Bronchoscopy in University Kebangsaan Malaysia Medical Centre (UKMMC).
Brief Title: Patient Satisfaction and Tolerability Using Virtual Reality (VR) as Adjunctive Treatment During Flexible Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Mohamed Faisal Abdul Hamid, Associate Professor, National University of Malaysia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ff-2021-506
Record Dates: First submitted 2022-03-14; First posted 2022-04-22 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Flexible Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient undergoing Bronchoscopy without use of VR device (No Intervention): patients undergoing flexible bronchoscopy without the VR device on, they will be shown a video consisting of calming nature scene together with soothing instrumental music. Sedation will be given as per standard practice.
- Patient Undergoing Bronchoscopy with the use of VR device (Experimental): patients undergoing flexible bronchoscopy with the VR device on, they will be shown a video consisting of calming nature scene together with soothing instrumental music. Sedation will be given as per standard practice.
  Interventions: Device: Virtual Reality Device

INTERVENTIONS:
Device: Virtual Reality Device — A virtual reality headset is a heads-up display (HUD) that allows users to interact with simulated environments and experience a first-person view (FPV). VR headsets replace the user's natural environment with virtual reality content, such as a movie, a game or a pre-recorded 360-degree VR environment that allows the user to turn and look around, just as in the physical world. Patient undergoing bronchoscopy will be given the device before and during the procedure.
  Arms: Patient Undergoing Bronchoscopy with the use of VR device

SUMMARY:
Flexible bronchoscopy is an important procedure used worldwide in the diagnosis and treatment of the disease of the of the lungs and airways . Flexible bronchoscopy is an invasive procedure that is utilized to visualize the nasal passages, pharynx, larynx, vocal cords, and tracheal bronchial tree. It is utilized for both the diagnosis and treatment of lung disorders. The procedure may be performed in an endoscopy suite, the operating room, the emergency department, a radiology suite, or at the bedside in the ICU. Flexible bronchoscopy (FB) is a safe procedure widely used in the management of patients with respiratory diseases. FB has close to zero mortality, and major complications are also very rare. Besides being safe and accurate, the comfort of the patient during the procedure is of primary concern of the medical and endoscopy staff.

Flexible Bronchoscopy can be a frightening and painful experience for the patient. There is room to improve the management of pain during FB, as many patients experience pain despite the common use of premedication analgesics and sedatives. In addition, because.

these medications have side effects, including respiratory depression and cardiovascular instability, it would be useful to develop nonpharmacologic approaches to improving the patient experience with painful procedures. The use of less medication may speed recovery from the procedure and facilitate the timely discharge of patients from the hospital. Nonpharmacologic practices, such as guided imagery, hypnosis, and distraction, have been effective in improving patient experiences during stressful or painful medical procedures. Distraction therapy is a technique in which sensory stimuli are provided to patients in order to divert their attention from an unpleasant experience. The use of nature scenes and sounds is an effective tool for distraction and has been successful in a variety of patient settings, including perioperative care, phlebotomy, and burn care. The benefit of nonpharmacologic approaches to analgesia during FB, however, has not been evaluated adequately. A visual reality (VR) device is an apparatus with a head up display (HUD) that projects a video and contains sound, the device is aimed to replace the patient's natural environment with virtual reality content. The use of Virtual reality(VR) device during flexible bronchoscopy has not been studies before.

DETAILED DESCRIPTION:
PROBLEM STATEMENT In Malaysia, flexible bronchoscopy has been well established in many respiratory centers as a means of diagnosis and treatment for many respiratory diseases, however there not many studies into use of nonpharmacological methods of improving patients experience during bronchoscopy. The use of conventional analgesia and sedation is considered standard of care during flexible bronchoscopy. In Respiratory centers, and our own center, Pusat Perubatan UKM (PPUKM), bronchoscopists use fentanyl and midazolam routinely as a means of analgesia during flexible bronchoscopy. There has not been research into the use of Virtual reality (VR) as a method of distraction to reduce anxiety and improve satisfaction in patient undergoing bronchoscopy. Investigators aim to carry out a randomize control trial, to study and compare the use Virtual Reality (VR) device in subjects undergoing flexible bronchoscopy. There are many parameters which the investigators will be looking into, the first will be overall subject's satisfaction with bronchoscope. Investigators will also compare parameter such as anxiety levels during the procedure, pain, cough and also breathlessness.

RESEARCH QUESTION Can VR (Virtual reality) device be used to improve satisfaction, reduce anxiety, pain cough and breathlessness for patients undergoing flexible bronchoscopy

HYPOTHESIS VR device can improve patient's satisfaction of flexible bronchoscopy by using methods of distraction.

VR device can reduce patient's anxiety during flexible bronchoscopy. VR device can reduce patient's pain during flexible bronchoscopy. VR device can reduce patient's cough during flexible bronchoscopy. VR device can reduce patient's breathlessness during flexible bronchoscopy.

OBJECTIVE General To compare satisfaction and tolerability of patients undergoing flexible bronchoscopy with or without VR (virtual reality).

Specific To compare pain score between patients with or without VR (virtual reality) before and after flexible bronchoscopy To compare Breathlessness score between patient with or without VR (virtual reality) before and after flexible bronchoscopy To compare severity of cough between patient with or without VR (virtual reality) before and after flexible bronchoscopy To compare anxiety between patient with or without VR (virtual reality) before and after flexible bronchoscopy

SIGNIFICANCE OF RESEARCH To determine new methods of audio-visual distraction as a method to increase patient satisfaction and tolerability of flexible bronchoscopy.

To determine if VR is a suitable to be used in the future for all patient undergoing Flexible Bronchoscopy.

This is a prospective interventional study conducted on patients undergoing flexible bronchoscopy under the Respiratory Unit, Department of Internal Medicine in UKMMC, who qualified both the inclusion and exclusion criteria. All eligible patients will be briefed about this study. Subsequently, consent will be obtained from those who are agreeing to participate, from the patient him/herself. The process of briefing and obtaining consent will be done prior to bronchoscopy when patient is in the waiting room. The patient will be randomized into 2 groups by block randomization 1:1(simple randomization), one undergoing flexible bronchoscopy with the VR device on, they will be shown a video consisting of calming nature scene together with soothing instrumental music. The other groups will undergo bronchoscopy without any device on Both groups will be given a questionnaire to assess pain, dyspnea and cough using a 10-point Visual analogue scale (VAS), ranging from 0 (no bother) to 10 (worst intolerable level) to determine a pre procedural baseline. Both groups of patients will be given the same amounts of sedation of midazolam 1 to 2 mg, with a supplemental 1-2mg midazolam and titrating dose of fentanyl from 12.5mg upwards. The interventional arm will be given the VR device to be worn 10 minutes before the procedure and will continue until the procedure is completed. Both groups of patients will be given another VAS questionnaire to assess pain, dyspnea, and cough during the procedure. The patient will also be given the State Trait Anxiety Inventory (STAI) questionnaire together with a satisfaction questionnaire, all of which to be answered 24 hours after the procedure to minimize any potential amnestic effect of the sedation given. The questionnaire and collection of data will not in any way interfere with the bronchoscopy procedure. Both groups with not differ in terms of standard of care during bronchoscopy. The VR device will be sanitized before every use using alcohol wipes so that the risk of infection will be minimized and users will be given disposable hygiene cover.

Standard Operating Procedure for COVID-19, for bronchoscopy. Firstly for the patient: a. Triaging of patients before entering bronchoscopy suite to be performed by medical staff. b. Patient and/or caregiver to scan My Sejahtera/ fill up screening and declaration form c. Ensuring patients to wear face mask. d. Ensuring patients to sanitize their hands using provided hand sanitizer. e. Temperature check. f. Suspected COVID-19 patients are directed to designated COVID-19 screening area. g. Practice of physical distancing of at least 1 meter among patients. h. All patient planned for bronchoscopy should have a Covid-19 Rapid antigen test kit (RTK) or reserve transcriptase polymerase chair reaction (RT-PCR) done at least 24-78hrs before bronchoscopy.

For the Bronchoscopy staff: a. All patients undergoing aerosol generating procedure (AGP) require thorough clinical assessment and COVID-19 diagnostic tests via RT-PCR for nasopharyngeal/ throat swabs as per local hospital protocols. Screening for other type of operation to be done if necessary. b. Appropriate personal protective equipment (PPE) should be worn in the ward for examination or procedures as stated for outpatient services. c. endoscopy and bronchoscopy should not be performed during the COVID-19 pandemic unless there is an absolute need for it. d. Rigid and flexible scope should be done in a designated procedure room to limit exposure to other staffs and patients. e. Appropriate PPE is to be worn for all procedure. f. Non-disposable equipment used during this procedure should be appropriately wrapped and covered to avoid virus contaminations. g. Sterilization of instruments and equipment used during the procedure is done according to infection control protocol. Discard all disposables accordingly.

For Aerosol Generating Procedures (AGPs). a. All procedures and surgeries should be performed while observing appropriate protective measures (PPE) in line with universal airborne, droplet and contact precautions. b. Procedures to be performed in designated COVID-19 operating theatre (OT) and ideally with negative pressure OT. c. All patients undergoing AGP require thorough clinical assessment and COVID-19 diagnostic tests via RT-PCR for nasopharyngeal/ throat swabs as per local hospital protocols. COVID-19 test for other type of operation to be done if necessary. d. If patient is not intubated, a surgical mask should be offered to the patient to wear at all times.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old and above
* Patient undergoing flexible bronchoscopy.
* understand and able to give consent (understand English and Malay)
* patient will need a negative covid PCR test as per standard practic

Exclusion Criteria:

* Age < 18
* Unable to understand and give consent (does not understand English, Malay)
* Ventilated patient
* Patient who are not comfortable wearing VR device
* Patient who are unable to communicate (illiterate, hearing impairment, mute, blind, Memory impairment)
* Patient on other sedation other than midazolam/fentanyl
* Patient undergoing other invasive examination planned alongside bronchoscopy.
* Patient with earlier history of bronchoscopy
* Patient with cranial-facial deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
To compare satisfaction and tolerability of patients undergoing flexible bronchoscopy with or without VR (virtual reality) using questionnaire, (0 - not satisfied, 5 extremely satisfied) | 6 months
  Both groups of patients will be given the same amounts of sedation of midazolam 1 to 2 mg, with a supplemental 1-2mg midazolam and titrating dose of fentanyl from 12.5mg upwards. The interventional arm will be given the VR device to be worn 10 minutes before the procedure and will continue until the procedure is completed. Both groups of patients will be given satisfaction questionnaire to be answered 24 hours after the procedure to minimize any potential amnestic effect of the sedation given.

SECONDARY OUTCOMES:
to compare pain of patient undergoing flexible bronchoscopy with or without VR (virtual reality), using a 10-point Visual analogue scale (VAS), ranging from 0 (no bother) to 10 (worst intolerable level) | 6 months
  Both groups of patients will be given the same amounts of sedation of midazolam 1 to 2 mg, with a supplemental 1-2mg midazolam and titrating dose of fentanyl from 12.5mg upwards. The interventional arm will be given the VR device to be worn 10 minutes before the procedure and will continue until the procedure is completed. Both groups of patients will be given a Visual analog scale (VAS) pain scale before endoscopy and another to be answered 24 hours after the procedure to minimize any potential amnestic effect of the sedation given.
to compare cough of patient undergoing flexible bronchoscopy with or without VR (virtual reality),using a 10-point Visual analogue scale (VAS), ranging from 0 (no bother) to 10 (worst intolerable level) | 6 months
  Both groups of patients will be given the same amounts of sedation of midazolam 1 to 2 mg, with a supplemental 1-2mg midazolam and titrating dose of fentanyl from 12.5mg upwards. The interventional arm will be given the VR device to be worn 10 minutes before the procedure and will continue until the procedure is completed. Both groups of patients will be given a Visual analog scale (VAS) cough scale before endoscopy and another to be answered 24 hours after the procedure to minimize any potential amnestic effect of the sedation given.
to compare breathlessness of patient undergoing flexible bronchoscopy with or without VR (virtual reality),using a 10-point Visual analogue scale (VAS), ranging from 0 (no bother) to 10 (worst intolerable level) | 6 months
  Both groups of patients will be given the same amounts of sedation of midazolam 1 to 2 mg, with a supplemental 1-2mg midazolam and titrating dose of fentanyl from 12.5mg upwards. The interventional arm will be given the VR device to be worn 10 minutes before the procedure and will continue until the procedure is completed. Both groups of patients will be given a Visual analog scale (VAS) breathlessness scale before endoscopy and another to be answered 24 hours after the procedure to minimize any potential amnestic effect of the sedation given.
to compare anxiety of patient undergoing flexible bronchoscopy with or without VR using Stat Trait Anxiety Index (STAI) questionairre. | 6 months
  Both groups of patients will be given the same amounts of sedation of midazolam 1 to 2 mg, with a supplemental 1-2mg midazolam and titrating dose of fentanyl from 12.5mg upwards. The interventional arm will be given the VR device to be worn 10 minutes before the procedure and will continue until the procedure is completed. Both groups of patients will be given a Stat Trait Anxiety Index (STAI) questionnaire after endoscopy to be answered 24 hours after the procedure to minimize any potential amnestic effect of the sedation given.

CONTACTS AND LOCATIONS:
Locations (3):
- Malaysia (3):
  - University Kebangsaan Malaysia Medical Center, Bandar Tun Razak, Cheras
  - National University of Malaysia, Cheras, Kuala Lumpur
  - University Kebangsaan Malaysia Medical Centre, Cheras, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunay E, Baki ED, Kokulu S, Ulasli SS, Oz G, Akar O, Bagcioglu E, Unlu M. Impact of multimedia information on bronchoscopy procedure: is it really helpful? Ann Thorac Med. 2015 Jan-Mar;10(1):34-7. doi: 10.4103/1817-1737.146862. PMID 25593605
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341
- [Background] Ni YL, Lo YL, Lin TY, Fang YF, Kuo HP. Conscious sedation reduces patient discomfort and improves satisfaction in flexible bronchoscopy. Chang Gung Med J. 2010 Jul-Aug;33(4):443-52. PMID 20804674
- [Background] Diette GB, Lechtzin N, Haponik E, Devrotes A, Rubin HR. Distraction therapy with nature sights and sounds reduces pain during flexible bronchoscopy: a complementary approach to routine analgesia. Chest. 2003 Mar;123(3):941-8. doi: 10.1378/chest.123.3.941. PMID 12628899
- [Background] Prakash UB, Offord KP, Stubbs SE. Bronchoscopy in North America: the ACCP survey. Chest. 1991 Dec;100(6):1668-75. doi: 10.1378/chest.100.6.1668. PMID 1959412
- [Background] Lechtzin N, Rubin HR, Jenckes M, White P, Zhou LM, Thompson DA, Diette GB. Predictors of pain control in patients undergoing flexible bronchoscopy. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):440-5. doi: 10.1164/ajrccm.162.2.9910022. PMID 10934067
- [Background] Fulkerson WJ. Current concepts. Fiberoptic bronchoscopy. N Engl J Med. 1984 Aug 23;311(8):511-5. doi: 10.1056/NEJM198408233110806. No abstract available. PMID 6749209
- [Background] Hirose T, Okuda K, Ishida H, Sugiyama T, Kusumoto S, Nakashima M, Yamaoka T, Adachi M. Patient satisfaction with sedation for flexible bronchoscopy. Respirology. 2008 Sep;13(5):722-7. doi: 10.1111/j.1440-1843.2008.01311.x. Epub 2008 May 29. PMID 18513244
- [Background] Lang EV, Benotsch EG, Fick LJ, Lutgendorf S, Berbaum ML, Berbaum KS, Logan H, Spiegel D. Adjunctive non-pharmacological analgesia for invasive medical procedures: a randomised trial. Lancet. 2000 Apr 29;355(9214):1486-90. doi: 10.1016/S0140-6736(00)02162-0. PMID 10801169
- [Background] Tusek DL, Church JM, Strong SA, Grass JA, Fazio VW. Guided imagery: a significant advance in the care of patients undergoing elective colorectal surgery. Dis Colon Rectum. 1997 Feb;40(2):172-8. doi: 10.1007/BF02054983. PMID 9075752
- [Background] Fernandez E. A classification system of cognitive coping strategies for pain. Pain. 1986 Aug;26(2):141-151. doi: 10.1016/0304-3959(86)90070-9. PMID 3531980
- [Background] Miller AC, Hickman LC, Lemasters GK. A distraction technique for control of burn pain. J Burn Care Rehabil. 1992 Sep-Oct;13(5):576-80. doi: 10.1097/00004630-199209000-00012. PMID 1452593
- [Background] Rusy LM, Weisman SJ. Complementary therapies for acute pediatric pain management. Pediatr Clin North Am. 2000 Jun;47(3):589-99. doi: 10.1016/s0031-3955(05)70227-3. PMID 10835992
- [Background] Hoffman HG, Patterson DR, Carrougher GJ. Use of virtual reality for adjunctive treatment of adult burn pain during physical therapy: a controlled study. Clin J Pain. 2000 Sep;16(3):244-50. doi: 10.1097/00002508-200009000-00010. PMID 11014398
- [Background] Gershon J, Zimand E, Pickering M, Rothbaum BO, Hodges L. A pilot and feasibility study of virtual reality as a distraction for children with cancer. J Am Acad Child Adolesc Psychiatry. 2004 Oct;43(10):1243-9. doi: 10.1097/01.chi.0000135621.23145.05. PMID 15381891
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Casalini AG, Majori M, Anghinolfi M, Burlone E, D'Ippolito R, Toschi M, Pisi G, Barantani D, Ghasempour D, Monica M. Foreign body aspiration in adults and in children: advantages and consequences of a dedicated protocol in our 30-year experience. J Bronchology Interv Pulmonol. 2013 Oct;20(4):313-21. doi: 10.1097/LBR.0000000000000024. PMID 24162114
- [Background] De S. Assessment of patient satisfaction and lidocaine requirement during flexible bronchoscopy without sedation. J Bronchology Interv Pulmonol. 2009 Jul;16(3):176-9. doi: 10.1097/LBR.0b013e3181afca25. PMID 23168547
- [Background] Cabrini L, Gioia L, Gemma M, Melloni G, Carretta A, Ciriaco P, Puglisi A. Acupuncture for diagnostic fiberoptic bronchoscopy: a prospective, randomized, placebo-controlled study. Am J Chin Med. 2006;34(3):409-15. doi: 10.1142/S0192415X06003941. PMID 16710890
- [Background] Jeppesen E, Pedersen CM, Larsen KR, Walsted ES, Rehl A, Ehrenreich J, Schnoor S, Backer V. Listening to music prior to bronchoscopy reduces anxiety - a randomised controlled trial. Eur Clin Respir J. 2019 Mar 17;6(1):1583517. doi: 10.1080/20018525.2019.1583517. eCollection 2019. PMID 30915199
- [Background] Triller N, Erzen D, Duh S, Petrinec Primozic M, Kosnik M. Music during bronchoscopic examination: the physiological effects. A randomized trial. Respiration. 2006;73(1):95-9. doi: 10.1159/000089818. Epub 2005 Nov 15. PMID 16293960
- [Background] Nilsson U. The anxiety- and pain-reducing effects of music interventions: a systematic review. AORN J. 2008 Apr;87(4):780-807. doi: 10.1016/j.aorn.2007.09.013. PMID 18395022
- [Background] Navidian A, Moulaei N, Ebrahimi Tabas E, Solaymani S. The effect of audiovisual distraction on the tolerability of flexible bronchoscopy: a randomized trial. Clin Respir J. 2018 Jan;12(1):76-83. doi: 10.1111/crj.12486. Epub 2016 May 10. PMID 27116084
- [Background] Garrett B, Taverner T, Gromala D, Tao G, Cordingley E, Sun C. Virtual Reality Clinical Research: Promises and Challenges. JMIR Serious Games. 2018 Oct 17;6(4):e10839. doi: 10.2196/10839. PMID 30333096